CLINICAL TRIAL: NCT06277830
Title: Wearable Sensor and Digital Technologies for Quantitative Assessment and Remote Monitoring of Symptoms in Myasthenia Gravis
Brief Title: Physical Activity Monitoring in Myasthenia Gravis
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: BioSensics (Industry)
Responsible Party: Principal Investigator, Amanda C. Guidon, MD, MPH, Assistant Professor of Neurology/Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 2023P002788
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Myasthenia Gravis
Keywords: telemedicine; wearable sensors; outcome measures; digital health; biomarkers; clinical trials
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adults with autoimmune myasthenia gravis: Existing patients at MassGeneral Hospital's MG clinic, ages 18-80, with autoimmune, AChR or MuSK antibody positive generalized myasthenia gravis.
  Interventions: Device: Wearable sensor

INTERVENTIONS:
Device: Wearable sensor — Participants will wear a pendant sensor for 7 days and then participate in an on-site examination with using a tablet designed to evaluate weakness in MG.
  Other Names: Tablet-based physical examination

SUMMARY:
The goal of this observational study is to evaluate the feasibility of using wearable sensor and digital technologies to measure motor and speech function in adults with autoimmune Myasthenia Gravis (MG).

The main question[s] it aims to answer are:

* To measure the correlation of sensor-based measures of motor function with existing outcome measures including the MG-ADL, MGQOL15r, QMG, MGComposite, and Neuro-QOL Fatigue scales.
* To develop and validate tablet-based digital assessments of speech and facial expression and to compare with existing outcome measures.

Participants will wear a pendant sensor for 7 days and then participate in tablet-based and in-person myasthenia-specific physical examinations. This will be performed in concert with routine care in the Massachusetts General Hospital MG clinic.

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is a chronic autoimmune neuromuscular disease characterized by fluctuating muscle weakness and symptoms that interfere with activities of daily living and negatively impacts quality of life. MG symptoms are currently assessed in person through a careful history and physical exam by a neuromuscular disease expert. Such in-clinic assessments are time-consuming, subjective, only provide a snapshot of a patient's disease and do not adequately reflect the spectrum of fluctuating weakness and symptoms. In 2019, NIH funded a rare disease clinical research consortium called MGNet. The consortium is focused on improved characterization of clinical phenotypes, discovery of biomarkers, and advancing clinical trial readiness for MG, which would enhance the development of more effective and personalized treatments. In this Fast Track SBIR project, BioSensics will collaborate with Massachusetts General Hospital - one of the key Consortium sites for MGNet - to develop and validate a wearable sensor solution (MGWear) for continuous remote monitoring of motor symptoms and function in MG patients and also a secure mobile application (MG app) for automatic assessment of speech and facial characteristics. The mobile application will also enable the transfer of data from the wearable device to BioSensics HIPAA-compliant backend cloud called BioDigit Cloud.

The objective of the study is to evaluate the feasibility of using wearable sensor and digital technologies to measure motor and speech function as well as developing metrics to measure ocular and facial expression to monitor disease activity and fluctuating muscle weakness in people with Myasthenia Gravis (MG).To achieve this objective, the investigators will conduct an observational study is to investigate the correlation between outcomes as measured by the PAMSys sensor and digital health technologies with the total score and sub-scores of MG specific outcome measures.

A key application and market for the proposed solution technology is pharmaceutical clinical trials. Wearable sensors and digital technologies like the technology proposed here could allow drug developers to test and iterate faster, providing a valuable new method for evaluating efficacy. Clinically, the proposed solution could be used to predict an individual's response to immunosuppressive drugs and to improve medication titration. Such solutions can enable detecting subtle changes in movement-based and digital biomarkers and provide insight into the phase of clinical disease onset. Additionally, the growing use of telemedicine to expand access and potentially reduce costs of high-quality care will require remote assessment strategies. 20% of states in the US (10 out of 50 states) have no specialized care for MG. Travel time, distance and cost may limit patients' access to expert care, even in states with identified MG specialists. The proposed remote monitoring technologies have potential to lessen barriers to quality care access for MG patients.

ELIGIBILITY:
Inclusion Criteria:

* Autoimmune generalized MG with or without history of thymoma, MGFA severity Class Ila/b, Illa/b or IVa
* Acetylcholine receptor antibody (AChR Ab) or muscle specific kinase receptor antibody (MuSK Ab) positive.
* Able to provide informed consent (physically/cognitively) and adhere with the protocol based on investigator's judgement
* Ambulatory, defined as able to independently walk a distance of 10 meters, with or without assistive device
* Male or female, aged 18-80 years
* Speaks English as primary language

Exclusion Criteria:

* Inability to engage in activities that are essential for independent living, such as dressing, bathing, toileting, eating independently.
* Neurological or orthopedic problems independent of myasthenia which significantly affects gait in the investigator's judgement
* Any significant medical, laboratory, or psychiatric condition that, in the judgment of the investigators, would potentially interfere with the ability to participate in the study
* Residence in long-term care centers or institutions, nursing facilities, skilled nursing facilities, or recipients of hospice care, or incarceration
* MGFA severity class IVb (severe bulbar weakness) or V (MG crisis)
* Pregnant or breastfeeding women
* Concurrent participation in an interventional clinical trial (observational studies, biomarker studies and registries are acceptable)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with generalized autoimmune myasthenia gravis who are existing patients in the Mass General Hospital Neuromuscular Clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | 1 week
  To measure the correlation of sensor-based measures of motor function to the MG-ADL, QMG, MGC, and Neuro-QOL Fatigue.

SECONDARY OUTCOMES:
Exploratory outcome | 1 week
  To develop and validate digital assessment of speech and facial expression compared to rating of MG-ADL, QMG, MGC, and Neuro-QOL Fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda C Guidon, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No